CLINICAL TRIAL: NCT00129207
Title: Effect of Ketoconazole Administration on the Pharmacokinetics and Pharmacodynamics of Bortezomib in Patients With Advanced Solid Tumors
Brief Title: Ketoconazole Administration: How it is Affected by the Body and Broken Down and How it Acts on the Body When Used With Velcade
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M34103-059
Record Dates: First submitted 2005-08-09; First posted 2005-08-11 (Estimated); Last update posted 2008-02-11 (Estimated); Status verified 2008-02

CONDITIONS: Tumors
Keywords: pharmacokinetic; pharmacodynamics; VELCADE; Ketoconazole; CYP 3A4; Solid Tumor; Advanced Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — Bortezomib

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
The purpose of this study is to investigate how ketoconazole (Nizoral) affects the pharmacokinetics (how the study drug is affected by the body and broken down) and pharmacodynamics (how the study drug acts on the body) of the active ingredient in the study drug Velcade (bortezomib).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 years of age or older, with a diagnosis of advanced solid tumor for which no curative or other treatment of higher priority is available
* Karnofsky Performance Status (KPS) equal to or greater than 70%
* Normal liver function tests (aspartate transaminase [AST] or alanine transaminase [ALT] equal to or less than 2 x upper limit of normal [ULN])
* Total bilirubin equal to or less than 1.5 x ULN
* Calculated creatinine clearance equal to or greater than 50 mL/min
* Normal serum calcium

Exclusion Criteria:

* Patients with significant cardiac disease
* Equal to or greater than Grade 2 neuropathy
* Active hepatitis
* HIV infection
* Secondary malignancy
* Transfusion-dependent or received extensive radiation therapy, systemic chemotherapy, or other antineoplastic therapy within 4 weeks of enrollment
* Patients taking concomitant medications having inhibitory or inducing activity for CYP 3A4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Primary Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center, UPMC Cancer Pavilion, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Venkatakrishnan K, Rader M, Ramanathan RK, Ramalingam S, Chen E, Riordan W, Trepicchio W, Cooper M, Karol M, von Moltke L, Neuwirth R, Egorin M, Chatta G. Effect of the CYP3A inhibitor ketoconazole on the pharmacokinetics and pharmacodynamics of bortezomib in patients with advanced solid tumors: a prospective, multicenter, open-label, randomized, two-way crossover drug-drug interaction study. Clin Ther. 2009;31 Pt 2:2444-58. doi: 10.1016/j.clinthera.2009.11.012. PMID 20110052